CLINICAL TRIAL: NCT01853462
Title: Effects of Supervised Balance and Proprioceptive Neuromuscular Facilitation Training After Lateral Ligament Sprains of the Ankle
Brief Title: Effects of Two Supervised Training Programs for the Rehabilitation of Ankle Sprains
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lazaros Lazarou (Other)
Responsible Party: Sponsor-Investigator, Lazaros Lazarou, Physiotherapist (MSc), Aristotle University Of Thessaloniki
Organization: Aristotle University Of Thessaloniki (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PNF-123-BAL-SPR
Record Dates: First submitted 2013-05-09; First posted 2013-05-15 (Estimated); Results first posted 2018-11-01 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-03

CONDITIONS: Ankle Sprains
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Proprioceptive Neuromuscular Facilitation (PNF) (Experimental): Supervised PNF training
  Interventions: Other: PNF training
- Balance (Experimental): Supervised balance training
  Interventions: Other: Balance training

INTERVENTIONS:
Other: PNF training — Ten individual PNF sessions, supervised by a physical therapist, with 50-60 min duration per session, within a maximal five-week period
  Arms: Proprioceptive Neuromuscular Facilitation (PNF)
Other: Balance training — Ten individual balance sessions, supervised by a physical therapist, with 50-60 min duration per session, within a maximal five-week period
  Arms: Balance

SUMMARY:
The purpose of this study was to determine the effects of supervised balance and proprioceptive neuromuscular facilitation (PNF) training for the rehabilitation of ankle sprains

DETAILED DESCRIPTION:
Supervised proprioceptive training has been recommended by recently published guidelines for the rehabilitation of ankle sprains. However, research evidence on the efficacy of this type of training is still weak, mainly owing to the methodological limitations of relevant studies. In addition, there is paucity of evidence concerning the effects of such training for the outcomes of functional performance, pain, ankle range of motion, and contradictory results have been reported for postural control.

This study aimed to substantiate the benefits of supervised training for the rehabilitation of ankle sprains, and elucidate the effects of two different proprioceptive protocols on the above-mentioned outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a symptomatic, conventionally treated, post acute (after 14 days) lateral ankle sprain, Grade I-II

Exclusion Criteria:

* Individuals with lateral ankle sprains Grade III
* Individuals with ankle sprain to the medial ligaments
* Individuals with ankle sprain to the interosseous (syndesmotic) ligament
* Individuals with concurrent fracture
* Individuals with chronic ankle instability
* Individuals with history of surgery to the ankles
* Individuals with history of lower limb nerve injuries
* Individuals with history of further ankle injuries, after the sprain
* Individuals with any injuries that hindered training participation

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2014-12; Primary Completion 2015-11 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lazaros S Lazarou, BSc, MSc, Principal Investigator — AristotleUniversity
Locations (1):
- Aristotle University, Serres, Agios Ioannis, Greece

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will be available only if necessarily required

RESULTS

PARTICIPANT FLOW:
Groups:
- Proprioceptive Neuromuscular Facilitation (PNF): PNF training
  proprioceptive neuromuscular facilitation exercise program: Ten individual sessions (50-60min per session) of PNF training, supervised by a physical therapist
- Balance: Balance training
  balance exercise program: Ten individual sessions (50-60min per session) of balance training, supervised by a physical therapist
Period: Overall Study
Arm/Group | Proprioceptive Neuromuscular Facilitation (PNF) | Balance
Started | 11 | 11
Completed | 10 | 10
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Proprioceptive Neuromuscular Facilitation (PNF) | Balance | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.8 (3.8) | 21.5 (1.8) | 21.7 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Ankle Functional Stability, Via the Single-leg Hop for Distance Test
Description: Participants hopped, using the sprained leg, as far forward as possible, and remained in the landing position for 2sec. Three trials were performed, and the mean hopping distance was used for analysis.
Time Frame: Baseline, after the completion of training (follow-up 1), and eight weeks after the completion of training (follow-up 2)
Measure: Mean (Standard Deviation); unit: Centimeters
Groups:
- Proprioceptive Neuromuscular Facilitation (PNF): Supervised Proprioceptive Neuromuscular Facilitation (PNF) Training
Arm/Group | Proprioceptive Neuromuscular Facilitation (PNF) | Balance
Number analyzed (Participants) | 10 | 10
Centimeters
  Baseline | 65.6 (17.0) | 82.8 (19.5)
  Follow-up 1 | 100.3 (17.0) | 101.4 (29.8)
  Follow-up 2 | 77.0 (17.6) | 110.0 (30.5)

2. Primary Outcome: Ankle Functional Stability, Via the Single-leg Hops for Time Test
Description: Participants hopped, using the sprained leg, as fast as possible, a six-meter distance. Three trials were performed, and the mean hopping time was used for analysis.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Proprioceptive Neuromuscular Facilitation (PNF) | Balance
Number analyzed (Participants) | 10 | 10
Seconds
  Baseline | 2.9 (0.6) | 3.3 (0.4)
  Follow-up 1 | 2.1 (0.2) | 2.7 (0.4)
  Follow-up 2 | 2.1 (0.3) | 2.2 (0.4)

3. Primary Outcome: Endurance of Ankle Dorsiflexor Muscles
Description: The rising on heel test was used, and participants rose on the heel of the sprained leg, as many times as possible.
  Scoring:10 points for >40 rises, 5 points for 30-39 rises, 0 points for <30 rises.
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: points on a scale
Arm/Group | Proprioceptive Neuromuscular Facilitation (PNF) | Balance
Number analyzed (Participants) | 10 | 10
points on a scale
  Baseline | 0 [0 to 10] | 5 [0 to 10]
  Follow-up 1 | 10 [5 to 10] | 10 [5 to 10]
  Follow-up 2 | 7.5 [0 to 10] | 10 [5 to 10]

4. Primary Outcome: Endurance of Ankle Plantar Flexor Muscles
Description: The rising on toes test was used, and participants rose on the toes of the sprained leg, as many times as possible. Scoring:10 points for >40 rises, 5 points for 30-39 rises, 0 points for <30 rises.
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: points on a scale
Arm/Group | Proprioceptive Neuromuscular Facilitation (PNF) | Balance
Number analyzed (Participants) | 10 | 10
points on a scale
  Baseline | 0 [0 to 0] | 0 [0 to 0]
  Follow-up 1 | 5 [0 to 10] | 7.5 [0 to 10]
  Follow-up 2 | 7.5 [0 to 10] | 7.5 [0 to 10]

5. Secondary Outcome: Anterior-posterior Stability Index
Description: The Biodex Stability System, which is a dynamic tilting platform, was used for assessment. The anterior-posterior stability index corresponded to the variance of foot platform displacement in the sagittal plane, and it was measured in single-leg stance, for the sprained leg, without footwear. Three 20-sec trials were performed, with open eyes, and the mean score was used for analysis.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Proprioceptive Neuromuscular Facilitation (PNF) | Balance
Number analyzed (Participants) | 10 | 10
Degrees
  Baseline | 2.6 (0.6) | 3.1 (0.6)
  Follow-up 1 | 2.6 (0.3) | 3.0 (0.7)
  Follow-up 2 | 2.5 (0.4) | 3.1 (0.7)

6. Secondary Outcome: Medial-lateral Stability Index
Description: The Biodex Stability System, which is a dynamic tilting platform, was used for assessment. The medial-lateral stability index corresponded to the variance of foot platform displacement in the frontal plane, and it was measured in single-leg stance, for the sprained leg, without footwear. Three 20-sec trials were performed, with open eyes, and the mean score was used for analysis.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Proprioceptive Neuromuscular Facilitation (PNF) | Balance
Number analyzed (Participants) | 10 | 10
Degrees
  Baseline | 1.9 (0.5) | 1.9 (0.4)
  Follow-up 1 | 1.7 (0.5) | 2.0 (0.5)
  Follow-up 2 | 1.6 (0.4) | 1.5 (0.3)

7. Secondary Outcome: Overall Stability Index
Description: The Biodex Stability System, which is a dynamic tilting platform, was used for assessment. The overall stability index corresponded to the variance of foot platform overall displacement, and it was measured in single-leg stance, for the sprained leg, without footwear. Three 20-sec trials were performed, with open eyes, and the mean score was used for analysis.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Proprioceptive Neuromuscular Facilitation (PNF) | Balance
Number analyzed (Participants) | 10 | 10
Degrees
  Baseline | 3.1 (0.7) | 3.6 (0.8)
  Follow-up 1 | 3.0 (0.6) | 3.4 (0.5)
  Follow-up 2 | 2.9 (0.6) | 3.4 (0.6)

8. Secondary Outcome: Ankle Dorsiflexion Range of Motion
Description: Assessement was performed with a goniometer. Participants actively dorsiflexed the sprained ankle, while being in long sitting, on a physical therapy table. The mean score of three measurements was used for analysis.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Proprioceptive Neuromuscular Facilitation (PNF) | Balance
Number analyzed (Participants) | 10 | 10
Degrees
  Baseline | 7 (3) | 8 (2)
  Follow-up 1 | 13 (3) | 15 (2)
  Follow-up 2 | 15 (2) | 15 (1)

9. Secondary Outcome: Pain Sensation
Description: The main component of the Greek version of the short form of McGill Pain Questionnaire (GR-SFMPQ) was used for the assessment of pain sensation of the sprained ankle. This consists of 15 descriptive adjectives for the pain sensation (11 sensory and 4 affective), which are self-rated according to their intensity level on a 4-point rating scale (0 = none, 1 = mild, 2 = moderate, 3 = severe). The total rating score (minimum = 0, maximum = 45) of the main component of the GR-SFMPQ was used for data analysis, with higher values representing a worse pain sensation.
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: Total score of scales
Arm/Group | Proprioceptive Neuromuscular Facilitation (PNF) | Balance
Number analyzed (Participants) | 10 | 10
Total score of scales
  Baseline | 7 [1 to 12] | 6 [2 to 10]
  Follow-up 1 | 0 [0 to 2] | 0 [0 to 2]
  Follow-up 2 | 3.5 [0 to 10] | 0.5 [0 to 1]

10. Secondary Outcome: Pain Intensity During the Week Before Testing
Description: The second component of the Greek version of the short form of McGill Pain Questionnaire, which is a visual analogue scale (VAS), was used for the assessment. The VAS is a horizontal 10-cm line with clearly defined boundaries: 0 cm = 'No pain' and 10.0 cm = 'worst possible pain'. partipants made a mark on the line at the point that better described the average pain intensity for their sprained ankle, during the week before testing. The distance marked from the 'no pain' point was measured in mm and was used for data analysis.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | Proprioceptive Neuromuscular Facilitation (PNF) | Balance
Number analyzed (Participants) | 10 | 10
Points on a scale
  Baseline | 2.0 (1.6) | 2.8 (2.1)
  Follow-up 1 | 0.4 (0.4) | 1.1 (1.3)
  Follow-up 2 | 1.3 (1.0) | 0.5 (0.7)

11. Secondary Outcome: Present Pain
Description: The third component of the Greek version of the short form of McGill Pain Questionnaire, which is a 6-point verbal rating scale, was used for the assessment. Participants noted what word at the time completing the questionnaire would best describe their pain sensation for the sprained ankle (scoring: no pain = 0, mild = 1, discomforting = 2, distressing = 3, horrible = 4, excruciating = 5). The score corresponding to the noted word was used for data analysis, with higher values representing a worse pain sensation.
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: Points on a scale
Arm/Group | Proprioceptive Neuromuscular Facilitation (PNF) | Balance
Number analyzed (Participants) | 10 | 10
Points on a scale
  Baseline | 1 [0 to 2] | 1 [0 to 2]
  Follow-up 1 | 0 [0 to 1] | 0 [0 to 1]
  Follow-up 2 | 1 [0 to 2] | 0 [0 to 1]

12. Secondary Outcome: Ankle Joint Sense for 10° Dorsiflexion
Description: The Biodex isokinetic dynamometer was used for assessment. During testing, participants were blindfolded, in the seated position, with footwear on.The internal goniometer of Biodex recorded the degrees of error for the active repositioning of 10° dorsiflexion (non-weight-bearing) for the sprained ankle, and the mean of three trials was used for analysis.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Proprioceptive Neuromuscular Facilitation (PNF) | Balance
Number analyzed (Participants) | 10 | 10
Degrees
  Baseline | 4 (2) | 6 (4)
  Follow-up 1 | 1 (1) | 3 (3)
  Follow-up 2 | 5 (3) | 4 (2)

13. Secondary Outcome: Ankle Joint Sense for 15° Plantar Flexion
Description: The Biodex isokinetic dynamometer was used for assessment. During testing, participants were blindfolded, in the seated position, with footwear on.The internal goniometer of Biodex recorded the degrees of error for the active repositioning of 15° plantar flexion (non-weight-bearing) for the sprained ankle, and the mean of three trials was used for analysis.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Proprioceptive Neuromuscular Facilitation (PNF) | Balance
Number analyzed (Participants) | 10 | 10
Degrees
  Baseline | 10 (4) | 9 (4)
  Follow-up 1 | 7 (3) | 5 (1)
  Follow-up 2 | 8 (3) | 5 (1)

14. Secondary Outcome: Ankle Joint Sense for 30° Plantar Flexion
Description: The Biodex isokinetic dynamometer was used for assessment. During testing, participants were blindfolded, in the seated position, with footwear on.The internal goniometer of Biodex recorded the degrees of error for the active repositioning of 30° plantar flexion (non-weight-bearing) for the sprained ankle, and the mean of three trials was used for analysis.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Proprioceptive Neuromuscular Facilitation (PNF) | Balance
Number analyzed (Participants) | 10 | 10
Degrees
  Baseline | 7 (6) | 4 (3)
  Follow-up 1 | 4 (2) | 3 (1)
  Follow-up 2 | 5 (2) | 3 (2)

15. Secondary Outcome: Peak Torque of Ankle Dorsiflexor Muscles at 30°/Sec Speed
Description: The Biodex isokinetic dynamometer was used for assessment. During isokinetic testing of the ankle joint, participants were in the seated position, with footwear on. Measurements were taken for the sprained leg, and the mean of five maximal trials was used for analysis.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Newton metres
Arm/Group | Proprioceptive Neuromuscular Facilitation (PNF) | Balance
Number analyzed (Participants) | 10 | 10
Newton metres
  Baseline | 35.8 (8.2) | 31.7 (6.8)
  Follow-up 1 | 30.7 (7.3) | 32.3 (8.6)
  Follow-up 2 | 30.8 (5.8) | 30.3 (7.3)

16. Secondary Outcome: Peak Torque of Ankle Dorsiflexor Muscles at 120°/Sec Speed
Description: as for outcome 15
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Newton metres
Arm/Group | Proprioceptive Neuromuscular Facilitation (PNF) | Balance
Number analyzed (Participants) | 10 | 10
Newton metres
  Baseline | 20.3 (4.2) | 22.7 (5.9)
  Follow-up 1 | 19.0 (5.4) | 21.4 (5.5)
  Follow-up 2 | 19.4 (4.1) | 22.1 (5.5)

17. Secondary Outcome: Peak Torque of Ankle Plantar Flexor Muscles at 30°/Sec Speed
Description: as for outcome 15
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Newton metres
Arm/Group | Proprioceptive Neuromuscular Facilitation (PNF) | Balance
Number analyzed (Participants) | 10 | 10
Newton metres
  Baseline | 31.5 (13.8) | 47.8 (23.6)
  Follow-up 1 | 46.1 (11.3) | 80.6 (31.4)
  Follow-up 2 | 53.5 (14.7) | 65.5 (25.5)

18. Secondary Outcome: Peak Torque of Ankle Plantar Flexor Muscles at 120°/Sec Speed
Description: as for outcome 15
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Newton metres
Arm/Group | Proprioceptive Neuromuscular Facilitation (PNF) | Balance
Number analyzed (Participants) | 10 | 10
Newton metres
  Baseline | 17.4 (4.6) | 26.0 (15.5)
  Follow up 1 | 25.0 (13.4) | 40.2 (12.1)
  Follow up 2 | 25.0 (8.6) | 38.1 (12.4)

19. Secondary Outcome: Peak Torque of Foot Evertor Muscles at 30°/Sec Speed
Description: The Biodex isokinetic dynamometer was used for assessment. During isokinetic testing of the subtalar joint, participants were in the seated position, with footwear on. Measurements were taken for the sprained leg, and the mean of five maximal trials was used for analysis.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Newton metres
Arm/Group | Proprioceptive Neuromuscular Facilitation (PNF) | Balance
Number analyzed (Participants) | 10 | 10
Newton metres
  Baseline | 11.9 (1.8) | 13.6 (2.5)
  Follow up 1 | 13.0 (3.8) | 14.5 (2.0)
  Follow up 2 | 13.9 (4.0) | 18.8 (2.3)

20. Secondary Outcome: Peak Torque of Foot Evertor Muscles at 120°/Sec Speed
Description: as for outcome 19
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Newton metres
Arm/Group | Proprioceptive Neuromuscular Facilitation (PNF) | Balance
Number analyzed (Participants) | 10 | 10
Newton metres
  Baseline | 8.0 (1.4) | 9.1 (1.5)
  Follow up 1 | 10.5 (2.3) | 8.6 (2.2)
  Follow up 2 | 10.5 (3.1) | 13.0 (3.0)

21. Secondary Outcome: Peak Torque of Foot Invertor Muscles at 30°/Sec Speed
Description: as for outcome 19
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Newton metres
Arm/Group | Proprioceptive Neuromuscular Facilitation (PNF) | Balance
Number analyzed (Participants) | 10 | 10
Newton metres
  Baseline | 10.1 (3.2) | 12.2 (3.8)
  Follow up 1 | 12.6 (5.6) | 18.6 (3.7)
  Follow up 2 | 26.2 (6.5) | 29.6 (9.9)

22. Secondary Outcome: Peak Torque of Foot Invertor Muscles at 120°/Sec Speed
Description: as for outcome 19
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Newton metres
Arm/Group | Proprioceptive Neuromuscular Facilitation (PNF) | Balance
Number analyzed (Participants) | 10 | 10
Newton metres
  Baseline | 6.7 (2.3) | 9.3 (3.5)
  Follow up 1 | 9.5 (3.2) | 12.0 (3.7)
  Follow up 2 | 21.6 (5.7) | 27.7 (8.9)

23. Secondary Outcome: Electromyographic Activity of Anterior Tibialis Muscle During Ankle Dorsiflexion at 30°/Sec Speed
Description: Two surface electrodes and a ground electrode were used for assessment. Measurements were taken for the sprained leg, during isokinetic testing of the ankle dorsiflexor muscles, at 30°/sec speed, with the Biodex dynamometer. Normalized values of the electromyographic (EMG) signals were used for analysis, and EMG activity during maximal voluntary isometric contraction of the anterior tibialis muscle was used as the reference value for normalization.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Proportion
Arm/Group | Proprioceptive Neuromuscular Facilitation (PNF) | Balance
Number analyzed (Participants) | 10 | 10
Proportion
  Baseline | 1.02 (0.25) | 0.88 (0.10)
  Follow up 1 | 0.90 (0.24) | 1.03 (0.10)
  Follow up 2 | 1.02 (0.27) | 0.92 (0.13)

24. Secondary Outcome: Electromyographic Activity of Anterior Tibialis Muscle During Ankle Dorsiflexion at 120°/Sec Speed
Description: Two surface electrodes and a ground electrode were used for assessment. Measurements were taken for the sprained leg, during isokinetic testing of the ankle dorsiflexor muscles, at 120°/sec speed, with the Biodex dynamometer. Normalized values of the electromyographic (EMG) signals were used for analysis, and EMG activity during maximal voluntary isometric contraction of the anterior tibialis muscle was used as the reference value for normalization.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Proportion
Arm/Group | Proprioceptive Neuromuscular Facilitation (PNF) | Balance
Number analyzed (Participants) | 10 | 10
Proportion
  Baseline | 0.99 (0.13) | 0.88 (0.23)
  Follow up 1 | 0.98 (0.17) | 0.85 (0.15)
  Follow up 2 | 1.02 (0.21) | 0.83 (0.13)

25. Secondary Outcome: Electromyographic Activity of Peroneus Longus Muscle During Ankle Plantar Flexion at 30°/Sec Speed
Description: Two surface electrodes and a ground electrode were used for assessment. Measurements were taken for the sprained leg, during isokinetic testing of the ankle plantar flexor muscles, at 30°/sec speed, with the Biodex dynamometer. Normalized values of the electromyographic (EMG) signals were used for analysis, and EMG activity during maximal voluntary isometric contraction of the peroneus longus muscle was used as the reference value for normalization.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Proportion
Arm/Group | Proprioceptive Neuromuscular Facilitation (PNF) | Balance
Number analyzed (Participants) | 10 | 10
Proportion
  Baseline | 0.78 (0.21) | 0.64 (0.09)
  Follow up 1 | 0.60 (0.16) | 0.76 (0.12)
  Follow up 2 | 0.61 (0.15) | 0.68 (0.14)

26. Secondary Outcome: Electromyographic Activity of Peroneus Longus Muscle During Ankle Plantar Flexion at 120°/Sec Speed
Description: Two surface electrodes and a ground electrode were used for assessment. Measurements were taken for the sprained leg, during isokinetic testing of the ankle plantar flexor muscles, at 120°/sec speed, with the Biodex dynamometer. Normalized values of the electromyographic (EMG) signals were used for analysis, and EMG activity during maximal voluntary isometric contraction of the peroneus longus muscle was used as the reference value for normalization.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Proportion
Arm/Group | Proprioceptive Neuromuscular Facilitation (PNF) | Balance
Number analyzed (Participants) | 10 | 10
Proportion
  Baseline | 0.82 (0.28) | 0.61 (0.15)
  Follow up 1 | 0.68 (0.21) | 0.71 (0.10)
  Follow up 2 | 0.71 (0.16) | 0.83 (0.12)

27. Secondary Outcome: Electromyographic Activity of Peroneus Longus Muscle During Foot Eversion at 30°/Sec Speed
Description: Two surface electrodes and a ground electrode were used for assessment. Measurements were taken for the sprained leg, during isokinetic testing of the foot evertor muscles, at 30°/sec speed, with the Biodex dynamometer. Normalized values of the electromyographic (EMG) signals were used for analysis, and EMG activity during maximal voluntary isometric contraction of the peroneus longus muscle was used as the reference value for normalization.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Proportion
Groups:
- Proprioceptive Neuromuscular Facilitation (PNF): Supervised Proprioceptive Neuromuscular Facilitation(PNF) Training
Arm/Group | Proprioceptive Neuromuscular Facilitation (PNF) | Balance
Number analyzed (Participants) | 10 | 10
Proportion
  Baseline | 0.89 (0.24) | 0.70 (0.22)
  Follow up 1 | 0.78 (0.22) | 0.68 (0.12)
  Follow up 2 | 0.92 (0.17) | 0.63 (0.16)

28. Secondary Outcome: Electromyographic Activity of Peroneus Longus Muscle During Foot Eversion at 120°/Sec Speed
Description: Two surface electrodes and a ground electrode were used for assessment. Measurements were taken for the sprained leg, during isokinetic testing of the foot evertor muscles, at 120°/sec speed, with the Biodex dynamometer. Normalized values of the electromyographic (EMG) signals were used for analysis, and EMG activity during maximal voluntary isometric contraction of the peroneus longus muscle was used as the reference value for normalization.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Proportion
Arm/Group | Proprioceptive Neuromuscular Facilitation (PNF) | Balance
Number analyzed (Participants) | 10 | 10
Proportion
  Baseline | 0.95 (0.34) | 0.75 (0.15)
  Follow up 1 | 0.67 (0.26) | 0.70 (0.15)
  Follow up 2 | 0.87 (0.43) | 0.74 (0.16)

29. Secondary Outcome: Electromyographic Activity of Tibialis Anterior Muscle During Foot Inversion at 30°/Sec Speed
Description: Two surface electrodes and a ground electrode were used for assessment. Measurements were taken for the sprained leg, during isokinetic testing of the foot invertor muscles, at 30°/sec speed, with the Biodex dynamometer. Normalized values of the electromyographic (EMG) signals were used for analysis, and EMG activity during maximal voluntary isometric contraction of the anterior tibialis muscle was used as the reference value for normalization.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Proportion
Arm/Group | Proprioceptive Neuromuscular Facilitation (PNF) | Balance
Number analyzed (Participants) | 10 | 10
Proportion
  Baseline | 0.40 (0.11) | 0.39 (0.10)
  Follow up 1 | 0.32 (0.13) | 0.40 (0.18)
  Follow up 2 | 0.54 (0.16) | 0.31 (0.15)

30. Secondary Outcome: Electromyographic Activity of Tibialis Anterior Muscle During Foot Inversion at 120°/Sec Speed
Description: Two surface electrodes and a ground electrode were used for assessment. Measurements were taken for the sprained leg, during isokinetic testing of the foot invertor muscles, at 120°/sec speed, with the Biodex dynamometer. Normalized values of the electromyographic (EMG) signals were used for analysis, and EMG activity during maximal voluntary isometric contraction of the anterior tibialis muscle was used as the reference value for normalization.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Proportion
Arm/Group | Proprioceptive Neuromuscular Facilitation (PNF) | Balance
Number analyzed (Participants) | 10 | 10
Proportion
  Baseline | 0.43 (0.12) | 0.44 (0.15)
  Follow up 1 | 0.45 (0.16) | 0.36 (0.14)
  Follow up 2 | 0.38 (0.14) | 0.32 (0.17)

31. Secondary Outcome: Participants With Recurrent Ankle Sprain
Time Frame: Twelve months after the completion of training
Measure: Count of Participants; unit: Participants
Arm/Group | Proprioceptive Neuromuscular Facilitation (PNF) | Balance
Number analyzed (Participants) | 10 | 10
Participants | 2 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data (not including serious) were collected during and after the completion of each individual training session
Description: The rating of perceived exertion was measured with the use of the Category Ratio-10 Borg Rating Scale. In addition, pain intensity was measured via a Numeric (0-10) Pain Rating Scale. For the measurements performed during training, participants who scored ≥4 ('somewhat strong' perceived exertion or more) in the Category Ratio-10 Borg Rating Scale or ≥5 ('moderate' pain or more) in the Numeric (0-10) Pain Rating Scale were free to interrupt training for that particular session.
Arm/Group | Proprioceptive Neuromuscular Facilitation (PNF) | Balance
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No